CLINICAL TRIAL: NCT05994404
Title: Cervical Spondylotic Myelopathy - Cost Observational Surgical Trial
Acronym: CSM-COST
Status: Completed | Type: Observational
Sponsor: Lahey Clinic (Other)
Collaborators: Mayo Clinic (Other)
Responsible Party: Sponsor
Other Study IDs: LCID: 2023; CE-1304-6173 (Other Grant/Funding Number: Patient-Centered Outcomes Research Institute)
Record Dates: First submitted 2023-07-28; First posted 2023-08-16 (Actual); Last update posted 2023-08-16 (Actual); Status verified 2023-07

CONDITIONS: Cervical Spondylosis With Myelopathy
Keywords: cost-effectiveness; cervical spondylotic myelopathy; health resource utilization; spinal fusion; laminoplasty

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Anterior Cervical Discectomy and Fusion: Ventral decompression and fusion was performed using multi-level discectomy (including partial or single level corpectomy) with fusion and plating. Allograft was used at each disc space and all compressive osteophytes were removed using the operating microscope. Plate fixation was done with rigid, semi-constrained, or dynamic titanium plates to optimize fusion and minimize complications.
  Interventions: Procedure: ACDF
- Posterior Instrumented Cervical Fusion: Dorsal decompression and instrumented fusion was performed using midline cervical laminoectom with the application of lateral mass screws and rods for rigid fixation. Local bone was used along with allograft to promote a lateral mass fusion.
  Interventions: Procedure: Posterior Cervical Fusion
- Laminoplasty: Laminoplasty was performed using an open-door approach with the application of plates and screws at each treated level. Ceramic or allograft laminar spacers (surgeon's choice) were used with titanium plates and screws to expand the spinal canal diameter.
  Interventions: Procedure: Cervical Laminoplasty

INTERVENTIONS:
Procedure: ACDF
  Groups: Anterior Cervical Discectomy and Fusion
Procedure: Posterior Cervical Fusion
  Groups: Posterior Instrumented Cervical Fusion
Procedure: Cervical Laminoplasty
  Groups: Laminoplasty

SUMMARY:
The purpose of the study is to determine the cost-effectiveness of different surgical strategies to treat cervical spondylotic myelopathy. The study will use data generated from the CSM-S Trial (NCT02076113).

1. To determine if laminoplasty is more cost-effective compared to dorsal fusion or ventral fusion surgery.
2. To determine the relative cost-effectiveness between anterior cervical discectomy and fusion (ACDF), posterior instrumented cervical fusion (PCF), and cervical laminoplasty.

DETAILED DESCRIPTION:
In this study, the investigators aim to cover a significant gap in the literature, namely, to compare anterior and posterior surgical approaches for the management of CSM on the cost of care. The investigators will conduct a post-hoc analysis of data from the randomized trial "Cervical Spondylotic Myelopathy Surgical Trial" (www.ClinicalTrials.gov; identifier: NCT02076113). This trial was conducted in collaboration between multiple academic institutions in North America. The results of the CSM-S RCT in terms of clinical and patient-reported outcomes suggested similar effectiveness with anterior and posterior surgical approaches. Notably, the study showed that cervical laminoplasty, a relatively low instrumentation-related cost procedure, was effective in managing CSM. The findings of the analysis proposed herein will add a new dimension to clinical decision-making by informing patient selection and improving the quality of care.

Post-hoc analysis will be conducted on the following data that were collected during the trial.

I. Functional outcomes determined by well-known quantitative scales (SF-36, Oswestry Neck, mJOA, and EuroQol-5D) at pre-op, 3 months, 6 months, 1 year, 2 years, 3 years, 4 years, and 5 years.

II. Health resource utilization information was collected using patient diaries along with copies of all medical bills and receipts at 1 month, 3 months, 6 months, and 12 months post-operatively for all patients. Participants were asked to monitor days missed from work and days unable to perform usual activities, in addition to days missed from work for medical treatments or evaluations.

The overall cost will be estimated for each patient from a societal perspective and will include the following components:

I. Index Hospitalization Cost - performed on all patients:

* Hospital Costs: Total hospital charges (TotalHC) will be used to estimate costs using hospital-specific and year-specific Medicare cost-to-charge ratios (CCR). The costs will be adjusted for inflation to the latest year of the study (2018) without a 3% discount. - Assumptions: cost-to-charge ratios for all hospitals and all relevant years will be provided. Data will be complete for all patients from all sites.

  o As a sub-analysis, hospital charges for specific revenue centers (i.e., radiology, pharmacy, physiotherapy, and occupational therapy) will be converted to costs using hospital-specific and year-specific CCRs. This will allow the identification of the major drivers of the difference in cost between the surgical strategies. A crosswalk between the revenue center and the cost center will have to be created. - Assumptions: Total hospital charges will be segmented out into the relevant revenue centers. All patients will have charges segmented in this manner. No major differences in how total hospital charges will be segmented by each site will exist.
* For professional services (identified with either HCPCS code or CPT-4 codes) provided to patients during the index hospitalization, costs will be calculated using national reimbursement amounts from the appropriate Medicare fee schedules for the respective year. - Assumptions: Detailed line-item services of all HCPCS codes and CPT-4 codes (including any necessary billing modifiers) will be provided for all professional services. Data will be complete for all patients from all sites.

II. One-year All-Cause Cost - performed on patients from sites capturing 1 year utilization:

• One-year all-cause costs will be calculated on hospital and professional services in the manner described above. - Assumptions: The same underlying assumptions described above.

III. Time to Return to Work - performed on all patients reporting employment:

* Investigators will assume that the work halted for patients on the procedure date).
* For patients to whom this outcome applies, the investigators will compare different cohorts using return to work as a time-to-event outcome.
* Lost wages will be estimated using the median weekly earnings in the US as reported by the Bureau of Labor Statistics.
* Patients providing no employment information will be assumed to have zero lost wages.
* Job-specific wages will not be estimated.

Index hospitalization costs and one-year all-cause costs will be combined with costs due to loss of productivity (indirect costs) to estimate total costs for each patient from a societal perspective. This will be performed on the subpopulation for which one-year costs were captured.

ELIGIBILITY:
Inclusion Criteria:

-Patients with Cervical Myelopathy (> or equal to 2 levels of spinal cord compression from C3 to C7) with 2 or more of the following symptoms/ signs: clumsy hands, gait disturbance, hyperreflexia, upgoing toes, bladder dysfunction.

Exclusion Criteria:

* C2-C7 kyphosis>5 degrees (measured in standing extension radiograph)
* segmental kyphotic deformity (defined by greater than 3 osteophytes extending dorsal to a C2-C7 dorsal-caudal line measured on cervical spine CT)
* structurally significant ossification of the posterior longitudinal ligament (OPLL - measured on cervical spine CT)
* previous cervical spine surgery, or significant active health-related co-morbidity (Anesthesia Class IV or higher)

Ages: 45 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study population consists of patients with multi-level cervical spondylotic myelopathy without kyphosis and who satisfied clinical equipoise criteria (ventral vs. dorsal approach) as judged by a panel of at least 15 spine experts.
Sampling Method: Non-Probability Sample
Enrollment: 269 (Actual)
Dates: Start 2014-04-01 (Actual); Primary Completion 2018-03-30 (Actual); Study Completion 2019-04-01 (Actual)

PRIMARY OUTCOMES:
Total Health Costs - Societal Perspective | 5 years
  Index hospitalization costs+one-year all cause costs+loss of productivity costs

SECONDARY OUTCOMES:
Index Hospitalization Costs | 30 days
  Hospital Costs
1-Year all-cause health costs | 1 year
  All health costs over 1 year
Loss of productivity costs | 5 years
  Costs associated with loss of productivity from a societal perspective

CONTACTS AND LOCATIONS:
Overall Officials: Zoher Ghogawala, MD, Study Director — Lahey Hospital & Medical Center; Robert G. Whitmore, MD, Principal Investigator — Lahey Hospital & Medical Center
Locations (2):
- United States (2):
  - Lahey Hospital & Medical Center, Burlington, Massachusetts
  - Mayo Clinic, Rochester, Minnesota

IPD SHARING:
Plan to Share IPD: Yes
De-identified data from the CSM-S trial including cost data will be available to other researchers who provide a valid study protocol.
Supporting Information: Study Protocol, SAP
Time Frame: Within 6 months of primary publication of the data and for 5 years thereafter
Access Criteria: Researchers with a clear and valid research protocol will be able to gain access to the data.

REFERENCES:
- [Result] Ghogawala Z, Terrin N, Dunbar MR, Breeze JL, Freund KM, Kanter AS, Mummaneni PV, Bisson EF, Barker FG 2nd, Schwartz JS, Harrop JS, Magge SN, Heary RF, Fehlings MG, Albert TJ, Arnold PM, Riew KD, Steinmetz MP, Wang MC, Whitmore RG, Heller JG, Benzel EC. Effect of Ventral vs Dorsal Spinal Surgery on Patient-Reported Physical Functioning in Patients With Cervical Spondylotic Myelopathy: A Randomized Clinical Trial. JAMA. 2021 Mar 9;325(10):942-951. doi: 10.1001/jama.2021.1233. PMID 33687463

DOCUMENTS (1):
  • Study Protocol (2023-07-10): https://cdn.clinicaltrials.gov/large-docs/04/NCT05994404/Prot_000.pdf